CLINICAL TRIAL: NCT01866059
Title: Randomised Controlled Clinical Trial to Compare Restorative Materials in the Treatment of Root Caries in an Older Irish Population.
Brief Title: Treatment of Root Caries in an Older Irish Population.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Martina Hayes, Clinical Research Fellow in Restorative Dentistry, University College Cork
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Root Caries Cork
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Active Root Caries; Over Sixty-five Years of Age; >=Two Carious Root Surfaces Per Patient
Keywords: root caries; GIC; RMGIC; Biodentine; Calcium silicate
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Calcium silicate cement (Experimental): Biodentine
  Interventions: Device: Calcium silicate cement
- Glass Ionomer Cement (Active Comparator): Fuji IX
  Interventions: Device: Glass Ionomer Cement
- Resin Modified Glass Ionomer Cement (Active Comparator): Fuji II LC
  Interventions: Device: Resin Modified Glass Ionomer Cement

INTERVENTIONS:
Device: Calcium silicate cement — Calcium silicate cement
  Other Names: Biodentine
  Arms: Calcium silicate cement
Device: Glass Ionomer Cement — Glass Ionomer Cement
  Other Names: Fuji IX
  Arms: Glass Ionomer Cement
Device: Resin Modified Glass Ionomer Cement — Resin Modified Glass Ionomer Cement
  Other Names: Fuji II LC
  Arms: Resin Modified Glass Ionomer Cement

SUMMARY:
This study will involve filling teeth which have decay on their roots with three different filling materials. Patients will attend Cork University Dental School and hospital for a clinical examination and to complete a questionnaire describing how they feel about the comfort and appearance of their teeth. Patients will be asked to provide a sample of saliva by spitting into a tube. This saliva will be tested to see what levels of bacteria are present and how well their saliva neutralises acid in their diet. This is used to assess how high or low the patient's risk of dental decay is. They will also complete a questionnaire about the amount of sugar in their diet and how often they clean their teeth. If the exam shows that any teeth are so decayed that they cannot be filled, the patient will then be offered extraction of these teeth. All treatment will be discussed with the patient. Patients will be randomly assigned one of the three materials and this material will be used for their fillings. Patients will not know which of the three materials they received but all three materials are already in use in dentistry and all of the elements of each treatment plan are well recognised, routine dental procedures. After all the treatment has been completed, each patient will be shown how best to take care of their teeth and how to manage their sugar intake to reduce their risk of further decay.

Patients will be given appointments to return for review at 6 months, 12 months, 18 months and 24 months after treatment. This will include a dental examination and dental impressions will be taken. These are used to measure how the restorative materials wear over time. Patients will also be asked to complete again the two questionnaires that they completed at their first visit to see if any of their answers have changed.

DETAILED DESCRIPTION:
Randomized Clinical Trial This study is a prospective study of older adults. It will assess the suitability of BiodentineTM as a filling material for Class V lesions and compare it's performance to that of Glass ionomer cement (GIC) and Resin-modified glass ionomer cement (RMGIC).

Patients for the study will attend Cork University Dental School and Hospital. These patients will represent a sample of the population of elderly who are generally well and able to care for themselves independently as well as adhere to a given maintenance programme. The general methods are outlined below.

Ethical Approval Ethical approval has been obtained from the Research Ethics Committee of the Cork Teaching Hospitals (CREC) for the recruitment, sampling, and treatment of elderly patients. Written informed consent will be obtained from all participants.

Inclusion Criteria

For inclusion in this research patients will:

* Be either male or female aged 65 or over
* Present a minimum of 6 teeth in one arch
* Have sufficient manual dexterity to undertake tooth-brushing
* Have sufficient cognitive ability to understand consent procedures and be able to complete a questionnaire

Exclusion Criteria

Patients will not be eligible for inclusion if:

* They are medically frail (ASA III or IV)
* They have pulpal involvement or painful symptomology other than sensitivity
* They have severe periodontal disease
* They require antibiotic prophylaxis for invasive dental treatment

Patient Recruitment (Phase 1) Prospective patients will be approached whilst attending Cork University Dental School and Hospital. General medical and dental practitioners in Cork will also be given information regarding the study to distribute to patients that may be suitable. A number of social clubs will also be approached. They will receive all the information in writing including the inclusion criteria as well as a consent form. If they indicate a willingness to participate, they will be offered an examination appointment. Insurance will be provided under the Clinical Indemnity Scheme, University College Cork.

Clinical Examination Procedure The clinical examination procedure will determine the extent of dental disease and confirm the suitability of the patient for enrolment in the study. Clinical data will be collected by a suitably trained examiner. This examiner will also provide the restorative treatment to the patients in the study.

During the course of the initial examination the following data will be collected:

* Age
* Gender
* Number of teeth
* Visually decayed, missing and filled teeth (VDMFT) index
* Visually decayed and filled root surfaces (RDFT)
* Plaque score
* Bleeding score
* Community Periodontal Index (CPI)
* Salivary flow rate
* Salivary buffer capacity (using CRT®buffer kits)
* Strep mutans count (using CRT®bacteria kits)
* Lactobacilli count (using CRT®bacteria kits)
* Denture wearing (Acrylic/Co-Cr, age of denture, abutment teeth)
* Fluoride exposure (public/private water supply, toothpaste, mouthwash)
* Medications (xerostomic potential, sucrose containing)
* Frequency of sugar intake
* Dental attendance pattern
* Alcohol consumption
* Smoking history
* Medical History
* Radiographs (where clinically indicated) The patient will be given another appointment to return if they are accepted into the trial.

Treatment Intervention (Phase 2) Each patient will be randomly assigned (using random number allocation) to be filled with one of three filling materials; Glass Ionomer Cement (GIC), Resin Modified Glass Ionomer Cement (RMGIC) and BiodentineTM. Treatment groups will be randomized and adjusted for the covariates age, gender and caries experience. Once it has been determined which filling material is to be placed in each lesion the treatment intervention stage will proceed as follows;

1. Scaling/prophylaxis to remove plaque and calculus
2. Removal of carious tissue from Class V lesions with hand or rotary instruments and restoration of the resulting cavities with the randomly assigned filling material

They will then be given review appointments for 6 months, one year, 18 months and two years. They will be sent appointment cards with the date of the next appointment by post and a phone call to confirm it.

Review Appointment (Phase 3) At each review appointment the following data will be gathered;

1. Survival and integrity of the restorations (according to USPHS Criteria)
2. Wear rates of the restorations (by means of dental impressions and contact profilometry)

Blinding A suitably trained examiner will assess the survival and integrity of the restorations placed by the principal investigator to eliminate potential bias.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 natural teeth with active root caries
* Aged 65 or older

Exclusion Criteria:

* Unable to give consent
* Edentulous
* No active carious root surfaces

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Survival of restorations | 2 year follow up
  Restorations will be assessed by a blinded examiner to determine whether they are still in situ or whether they have been lost.

CONTACTS AND LOCATIONS:
Overall Officials: Finbarr Allen, Principal Investigator — University College Cork; Martina Hayes, Principal Investigator — University College Cork; Frank Burke, Study Chair — University College Cork
Locations (1):
- Cork University Dental School and Hospital, Cork, Cork, Ireland

REFERENCES:
- [Derived] Hayes M, da Mata C, Tada S, Cole M, McKenna G, Burke FM, Allen PF. Evaluation of Biodentine in the Restoration of Root Caries: A Randomized Controlled Trial. JDR Clin Trans Res. 2016 Apr;1(1):51-58. doi: 10.1177/2380084416628474. PMID 30931695